CLINICAL TRIAL: NCT01253837
Title: Phase I/II Study of the Tumor-targeting Human L19TNFα Monoclonal Antibody-cytokine Fusion Protein in Patients With Advanced Solid Tumors
Brief Title: L19TNFα in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Philogen S.p.A. (Industry)
Collaborators: InnoPharma Inc. (Industry); Eudax S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-L19TNFα-02/07; 2007-001157-26 (EudraCT Number)
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Solid Tumors; Colorectal Cancer
Keywords: L19; antibody; monoclonal; tumor targeting; TNFa; colorectal cancer; Phase I: Patients with relapsed or refractory locally advanced or metastatic solid tumors not amenable to standard systemic therapy.; Phase II: Patients with relapsed or refractory locally advanced or metastatic colorectal cancer not amenable to standard systemic therapy.
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- L19TNFa (Experimental): Phase I: Prospective, open-label, dose escalation study.
  Phase II: Prospective, single-arm, open-label study, equivalent to the stage 1 of the Simon two-stage phase II design.
  Interventions: Drug: L19TNFa

INTERVENTIONS:
Drug: L19TNFa — Phase I: Sequential assignment of Patient cohorts to one of six dose levels of L19TNFa: 1.3, 2.6, 5.2, 7.8, 10.4, 13.0 µg/kg.
  Phase II: The Recommended Dose (RD) of 13.0 µg/kg of L19TNFα determined in Phase I.
  Schedule: Infusions of L19TNFα on days 1, 3 and 5 of each 21-day cycle. Patients may remain on treatment for a maximum of six 21-day cycles.

SUMMARY:
The recombinant human fusion protein L19TNFα was created with the intention to overcome the systemic toxicity of TNFα by directly targeting it to tumor tissues. Tumor-targeted L19TNFα would result in high and sustained intralesional bioactive TNFα concentrations.

DETAILED DESCRIPTION:
The primary purpose of this Phase I/II study is to define a safe and potentially active treatment regimen of L19TNFα as a monotherapy and to evaluate the antitumor activity of this regimen in relapsed metastatic colorectal cancer subjects, for whom standard treatment options are exhausted. L19TNFα is an investigational drug that specifically and effectively binds to ED-B, which is abundantly expressed in cancer tissue. Accordingly, treatment should result in a high and long-lasting intratumoral accumulation of biologically active rh-TNFα. Although combined therapies of TNFα with cytotoxic drugs (e.g. melphalan) seem to be strikingly more active against sarcoma and melanoma than with TNFα alone - at least for the ILP setting it seems possible that the repeated intratumoral delivery of TNFα via L19TNFα might produce additional biologic effects, such as the induction of an immunologic antitumor response or the sustained inhibition of tumor-associated angiogenesis (Lejeune, 2006), that potentially could benefit advanced cancer subjects.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: histologically or cytologically confirmed relapsed or refractory locally advanced or metastatic solid tumor of any origin, not amenable to standard therapy.
* Phase II: histologically or cytologically confirmed relapsed or refractory locally advanced or metastatic colorectal cancer not amenable to standard therapy.
* For both phase I and II:

  * Subjects aged ≥ 18 years.
  * ECOG performance status ≤ 2.
  * Subjects must have at least one unidimensionally measurable lesion by computed tomography as defined by RECIST criteria (see Section 8) or tumour markers parameters of disease such as PSA and CA125 for Prostate cancer and Ovarian cancer, respectively. This lesion must not have been irradiated during previous treatments.
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, platelets ≥ 100 x 10^9/L, and haemoglobin (Hb) ≥ 9.5 g/dl.
  * All acute adverse effects (excluding alopecia) of any prior therapy (including surgery, radiation therapy, chemotherapy) must have resolved to ≤ Grade 1, except elevated liver transaminases judged to be associated with tumor infiltration (see below) (graded according to National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events, version 3.0 [CTCAE, v.3.0]).
  * Alkaline phosphatase (ALP), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN), and total bilirubin ≤ 2.0 mg/gL unless liver involvement by the tumor, in which case the transaminase levels up to 5 x ULN are allowed.
  * Creatinine ≤ 1.5 ULN or 24 h creatinine clearance ≥ 60 mL/min.
  * Testing negative for acute or chronic infection with hepatitis B or C virus, or human immunodeficiency virus 1 or 2.
  * Negative pregnancy test for females of childbearing potential at the screening visit.
  * Commitment from subject to practice medically appropriate/acceptable method of birth control (e.g., hormonal, condoms or other adequate barrier controls, intrauterine contraceptive device, or sterilization) beginning at the screening visit and continuing until 3 months following the last treatment with study drug.
  * Able to provide written Informed Consent.

Exclusion Criteria:

* Breastfeeding women.
* Presence of active infections (e.g. requiring antimicrobial therapy) or other severe concurrent disease, which, in the opinion of the Investigator, would place the subject at undue risk or interfere with the study.
* Known brain metastases or signs and/or symptoms suggestive of brain metastases.
* Known cancer of other primary origin (excluding Stage I non-melanoma skin cancer) within the prior 5 years.
* Active autoimmune disease.
* Cardiac disease as manifested by any of the following:

  * > Grade II heart failure, graded per New York Heart Association (NYHA) criteria.
  * Unstable angina pectoris.
  * Acute or subacute coronary syndromes, including myocardial infarction, occurring with 1 year prior to study treatment.
  * Arrhythmia needing continuous treatment.
  * Ejection fraction less than the institutional lower limit of normal as assessed by multigated radionuclide angiography (MUGA) scan or echocardiogram.
* Uncontrolled hypertension.
* Ischemic peripheral vascular disease (Grade IIb-IV).
* Severe diabetic retinopathy.
* Major surgery or trauma within 4 weeks prior to start of study treatment.
* Known history of allergy to TNFα or other intravenously administered human proteins/peptides/antibodies.
* Chemotherapy, radiation therapy or therapy with an investigational agent within 4 weeks prior start of study treatment.
* Previous in vivo exposure to monoclonal antibodies for biological therapy in the 6 weeks before administration of study treatment.
* Growth factors or immunomodulatory agents within 7 days prior to the administration of the study treatment.
* Subject requires or is taking corticosteroids or other immunosuppressant drugs on a long-term basis. Limited use of corticosteroids to treat or prevent acute hypersensitivity reactions is not considered an exclusion criterion.
* Concurrent therapy with warfarin at doses greater than 1 mg/day or equivalent doses of other coumarin derivatives.
* Participation in another interventional clinical trial during participation in this trial.
* Expectation that the subject will not be able to complete at least 6 weeks of therapy.
* Any conditions that in the opinion of the Investigator could hamper compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2007-09; Primary Completion 2011-05 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Phase I: Determination of the Maximum Tolerated Dose (MTD) and Recommended Dose (RD) | day 1-29
  Determination of the Maximum Tolerated Dose (MTD) and Recommended Dose (RD) of L19TNFα.
Phase II: Investigation of the anti-cancer activity of L19TNFα as measured by Objective Response Rate (ORR) | within day 42
  Investigation of the anti-cancer activity of L19TNFα as monotherapy as measured by the Objective Response Rate (ORR) at the end of cycle 2 in subjects with relapsed or refractory locally advanced or metastatic colorectal cancer not amenable to standard systemic therapy.

SECONDARY OUTCOMES:
Investigation of serum concentrations of L19TNFα (pharmacokinetic properties) | day 1-5
Investigation of the induction of human anti-fusion protein antibody (HAFA) | 1-16 months
Investigation of early signs of anti-tumor activity of L19TNFα | 14 months
  Investigation of early signs of anti-tumor activity of L19TNFα as measured by Objective Response Rate (ORR) at the end of cycle 2, median Progression-Free Survival (PFS) and median Overall Survival (OS).

CONTACTS AND LOCATIONS:
Overall Officials: Filippo De Braud, Dr., Principal Investigator — European Istitute of Oncology Milan (Italy)
Locations (2):
- Italy (2):
  - A.O. UNIVERSITARIA OSPEDALI RIUNITI - OSPEDALE UMBERTO I DI ANCONA - ANCONA (Italy), Ancona
  - European Istitue of Oncology Milan (Italy), Milan